CLINICAL TRIAL: NCT02993991
Title: Pre-operative Mocetinostat (MGCD0103) and Durvalumab (MEDI4736) (PRIMED) for Squamous Cell Carcinoma of the Oral Cavity
Acronym: PRIMED-001
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated due to a change in internal prioritization and not due to any safety concerns.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mirati Therapeutics Inc. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIMED-001
Record Dates: First submitted 2016-12-01; First posted 2016-12-15 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Squamous Cell Carcinoma, Head And Neck; Squamous Cell Carcinoma Mouth; Resectable Squamous Cell Carcinoma of Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — mocetinostat; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mocetinostat and Durvalumab (Experimental): Patients will start therapy with mocetinostat within 10 days of study enrollment. Mocetinostat will be given in 2 dose levels (n = 6 evaluable patients each) of 70mg three-times weekly and 90mg three-times weekly for 2 weeks.
  Durvalumab will be given as a single infusion at a dose of 1500mg, over a period of 1-hour, on day 8 of the study.
  Interventions: Drug: Mocetinostat; Biological: Durvalumab

INTERVENTIONS:
Drug: Mocetinostat — Mocetinostat (MGCD0103) is a potent small molecule HDAC inhibitor that targets human HDAC isoforms. It is an orally bioavailable, second generation benzamide inhibitor of HDAC 1, 2, 3 and 11 with broad spectrum antitumor activity in vitro and in vivo.
  Other Names: MGCD0103
Biological: Durvalumab — Durvalumab is a human immunoglobulin G1 kappa (IgG1κ) monoclonal antibody directed against human PD-L1. It is selective for recombinant PD-L1 and blocks the binding of recombinant PD-L1 to the PD-1 and CD80 receptors.
  Other Names: MEDI4736

SUMMARY:
This is a Phase 1 Window of Opportunity study to evaluate the pharmacodynamic and immune effects of pre-operative therapy with Mocetinostat and Durvalumab on patients with squamous cell carcinoma of the oral cavity.

DETAILED DESCRIPTION:
This is a single center, open-label, non-randomized, pre-operative window of opportunity study for patients with resectable squamous cell carcinoma of the oral cavity who are considered suitable for curative-intent surgical resection, with pre-operative Mocetinostat and Durvalumab.

This study will involve treatment with Mocetinostat and Durvalumab, tests and procedures done for safety and the collection of blood samples for biomarker research. Tissue samples (fresh biopsy or archival tissue) will also be collected for biomarker research and evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written and voluntary informed consent.
2. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Age > 18 years, male or female. Disease characteristics
4. Patient must be diagnosed with histologically confirmed squamous cell carcinoma of the oral cavity (SCCOC) (floor of mouth, anterior 2/3 tongue, buccal mucosa, upper and lower gingiva, and retromolar trigone) considered resectable by the head and neck surgical rounds (T2-4a, N0-2, M0; without evidence of distant metastasis).
5. Patient must be willing and able to provide up to 2 fresh tumor biopsies for histopathological and biomarker evaluation; first as pre-treatment baseline, and the second after treatment with mocetinostat but prior to treatment with durvalumab.

   * Patients who decline an in-house fresh pre-treatment tumor biopsy must give consent to provide a tumor block from an existing diagnostic primary tumor biopsy completed within 90 days of enrollment, which is of acceptable quality and quantity for analysis, as assessed by the study site correlatives team.
6. No anti-neoplastic treatment is allowed between the time from obtaining baseline tumor specimen and enrollment.

   Patient characteristics
7. ECOG performance status 0-1.
8. Patient must have adequate organ function as determined by the following:

   - Renal function: i. Serum creatinine < 1.5 ULN (upper limit of normal range) or a calculated creatinine clearance of > 50mL/min using the following formula: Creatinine clearance = [(140-age) x wt (kg) x Constant*] / creatinine (umol/L)

   *Constant = 1.23 for men, and 1.04 for women

   - Bone marrow function (without hematopoietic growth factors or transfusion): i. Absolute neutrophil count (ANC) > 1.5 x 109/L ii. Leukocytes > 3.0 x 109/L iii. Hemoglobin > 90 g/L or > 9g/dL iv. Platelets > 100 x 109/L

   - Liver function: i. Total bilirubin < ULN ii. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < 2.5 x ULN

   - Cardiac function: i. A normal left ventricular ejection fraction (LVEF) of > 50% and the absence of any clinically significant pericardial effusion, as evidenced by an echocardiogram performed within 4 weeks of the study commencement.
9. Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
10. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Primary site of head and neck carcinoma unknown, lip, hard palate, skin, or outside the oral cavity.
2. Patients with tumors that invade major vessels, as shown unequivocally by imaging studies.

   * For patients with tumors that do not invade major blood vessels but are within 3mm of the carotid artery or branches thereof, any anticoagulant therapy (including aspirin, non-steroidal anti-inflammatories, antiplatelet agents or other anti-coagulants) must be discontinued.
3. Patients with any prior history of bleeding related to the current head and neck cancer.
4. Patients with a history of gross hemoptysis (bright red blood of ½ teaspoon or more per episode of coughing) < 3 months prior to enrollment.
5. Prior or concurrent radiation therapy to tumor at site of planned resection.
6. Any concurrent chemotherapy, biologic, immunologic or hormonal therapy for cancer treatment.

   * Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
7. Current or prior use of immunosuppressive medication within 14 days prior to starting dosing. The following are exceptions to this criteria:

   * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection).
   * Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent.
   * Steroids as premedication for hypersensitivity reactions (eg, computed tomography scan premedication).
8. Active or documented history of autoimmune disease within 2 years before screening, including:

   * Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis).
   * Patients with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, Grave's disease, Hashimoto's disease, or psoriasis not requiring systemic treatment within the past 2 years, are not excluded.
9. History of primary immune deficiency.
10. History of organ transplant that requires use of immunosuppressive medications.
11. Use of any live vaccines against infectious diseases within 4 weeks of study treatment initiation.
12. Known allergy or reaction to any component of Mocetinostat and/or Durvalumab formulation.
13. Known history of tuberculosis.
14. Subjects who are known to be human immunodeficiency (HIV) positive.
15. Subjects who are known to be hepatitis B or C positive.
16. Female patients who are pregnant or breast-feeding.
17. Male or female patients of reproductive potential who are not willing to use effective birth control from screening to 180 days following the last dose of durvalumab.
18. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, unstable cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events from Mocetinostat or Durvalumab, or compromise the ability of the subject to give written informed consent.
19. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results.
20. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
21. History of another primary malignancy, except for:

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence,
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease,
    * Adequately treated carcinoma in situ without evidence of disease.
22. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study medications.
23. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-10 (Estimated); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effects with biomarker analyses (Tumor PD-L1 by IHC; Density of peri-tumoral and intra-tumoral CD3, CD4 and CD8-positive lymphocytes; Serum pro-inflammatory cytokines and chemokines) | 3 years
Immune effects with biomarker analyses (Tumor PD-L1 by IHC; Density of peri-tumoral and intra-tumoral CD3, CD4 and CD8-positive lymphocytes; Serum pro-inflammatory cytokines and chemokines) | 3 years

SECONDARY OUTCOMES:
Toxicities as per NCI CTCAE v4.1 | 3 years
Rate of completion of surgery within the initially planned window as per RECIST v1.1 | 3 years
Rate of disease progression as per RECIST v1.1 during the pre-operative treatment period | 3 years
Rate of post-operative complications as per NCI CTCAE v4.1 | 3 years
Optimal biologically active dose of mocetinostat (Correlation of tumor and serum-based assessments with mocetinostat dose levels) | 3 years
Changes in serum mocetinostat concentrations prior to and following durvalumab therapy | 3 years

OTHER OUTCOMES:
Dynamic changes in immune cell activation and/or suppression using flow cytometry and DNA/RNA sequencing (tumor and immune cell genome and trascriptome analysis) | 3 years
Dynamic changes in intratumoral hypoxia with pre-operative mocetinostat and durvalumab therapy using 18FAZA PET | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Staff Physician and Medical Oncologist
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada